CLINICAL TRIAL: NCT01453790
Title: Effectiveness of Parent Specific Depression Education and Motivation on Intent to Seek Follow-Up Care for Potential Depression Symptoms
Brief Title: Parent Specific Depression Education and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 214808; 214808-7 (Other: UC Davis)
Record Dates: First submitted 2011-10-11; First posted 2011-10-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-06

CONDITIONS: Depressive Symptoms
Keywords: depression; treatment; motivation to seek follow up
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent-Specific Depression Education-Motivation (Experimental): Mothers receive depression education (verbal and written) with messages targeted to parent status which are drawn from previous research. They also receive motivational messages at 2 days via telephone.
  Interventions: Behavioral: Parent-Specific Depression Education and Motivation
- General Depression Education (Active Comparator): Mothers receive general depression education (verbal and written) which are drawn from previous research. They also receive attention control telephone calls at 2 days.
  Interventions: Behavioral: General Depression Education-Motivation

INTERVENTIONS:
Behavioral: Parent-Specific Depression Education and Motivation — Parent-specific written and verbal depression messages garnered from previous research were consolidated into a pamphlet and script, respectively. These are dispensed after randomization in the pediatric office. At two days, mothers in the experimental group receive a motivational telephone call.
  Arms: Parent-Specific Depression Education-Motivation
Behavioral: General Depression Education-Motivation — General depression education messages were compiled and are delivered verbally (scripted) and written (JAMA Depression Patient Page) after randomization in the pediatric office. At 2 days, mothers in the comparison group receive an attention control telephone call.
  Arms: General Depression Education

SUMMARY:
This project is an investigator-initiated, randomized-controlled trial of the effectiveness of written and verbal parent-specific depression education and motivational advice in increasing participants self-disclosed intention to seek follow-up care for possible depression symptoms. The control condition is written and verbal general depression education and advice. Hypothesis: the office-based experimental intervention of written and verbal parent-specific depression and emotional health education and motivational advice increases intention to seek follow-up services for emotional health or depression, when compared to written and verbal general depression education and advice.

DETAILED DESCRIPTION:
Maternal depression is a common problem, debilitating for mothers and affecting parenting practices with negative effects on the behavior, development, and physical health of children. The value of identifying and treating maternal depression for child development and well-being is well documented. Unfortunately, there are multiple barriers to the recognition and treatment of maternal depression. This is particularly problematic in younger women, as they are less often seen for health care. The overall objective of this project is to test whether the uptake of follow-up recommendations for potential depression by mothers identified by screening in clinical settings is improved by parent-specific targetting of depression education and motivational advice.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child between the ages of 2 days and 12 years who is a patient of the UC Davis Pediatric Clinic.
* Primary, female caregiver
* Feeling down, depressed, or hopeless or little interest or pleasure in doing things.
* Not currently receiving care from a mental health practitioner.
* Comfortable speaking English without an interpreter.

Exclusion Criteria:

* Parent of a child younger than 2 days or older than 12 years.
* Dad, Foster parent, or other short term guardian.
* Currently in treatment with a mental health practitioner.
* Limited English Proficiency

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Depression Follow-Up Care Seeking | at 2 weeks
  Mothers' self-reported attempts at obtaining follow-up services for emotional health or depression.

SECONDARY OUTCOMES:
Intention to Seek Depression Follow-Up Care | at 2 weeks
  Three item scale measure of intention to seek care (any) for follow-up of positive depression screen.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, General Pediatrics, Sacramento, California, United States

REFERENCES:
- [Derived] Fernandez y Garcia E, Joseph J, Wilson MD, Hinton L, Simon G, Ludman E, Scott F, Kravitz RL. Pediatric-based intervention to motivate mothers to seek follow-up for depression screens: The Motivating Our Mothers (MOM) trial. Acad Pediatr. 2015 May-Jun;15(3):311-8. doi: 10.1016/j.acap.2014.11.008. PMID 25906700